CLINICAL TRIAL: NCT01641796
Title: Paromomycin Topical Cream Treatment Protocol for Individuals With Uncomplicated Cutaneous Leishmaniasis
Brief Title: Paromomycin for Individuals With Uncomplicated Cutaneous Leishmaniasis
Status: No longer available | Type: Expanded Access
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: S-12-13; S-12-13/M-10337 (Other: The Surgeon General Department of the Army)
Record Dates: First submitted 2012-06-18; First posted 2012-07-17 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Leishmaniasis, Cutaneous
Keywords: Cutaneous Leishmaniasis; CL; Lesion; Topical; Treatment; Cream; Expanded Access
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Paromomycin

INTERVENTIONS:
Drug: Paromomycin — Paromomycin Topical Cream applied to all lesions once a day for 20 days
  Other Names: Paromomycin Topical Cream

SUMMARY:
This is an expanded access treatment protocol designed to provide a topical cream treatment option to military health care beneficiaries with parasitologically confirmed uncomplicated Cutaneous Leishmaniasis.

DETAILED DESCRIPTION:
When a military health care beneficiary presents at a Department of Defense Military Treatment Facility with a skin lesion clinically and epidemiologically consistent with suspicious Cutaneous Leishmaniasis (CL), routine diagnostic parasitology testing will be performed as standard of care, and if there is a positive diagnosis, the patient will be offered the option to participate in this treatment program and after providing written informed consent/assent., if eligible to participate, the patient will receive treatment with Paromomycin Topical Cream.

Eligible patients will receive Paromomycin Topical Cream applied topically to all CL lesions once daily for 20 days. The Day 1 application will be performed by or under the supervision of the site PI. The Day 2 application will be performed by the patient while being observed by the site PI or a designated medical staff member. The patient will be scheduled to return to an Medical Treatment Facility (MTF) weekly during treatment at Days 7 ± 2, 14 ± 2, and Day 20 + 4 days (the last day of treatment). During these visits, a member of the medical team will observe the application of the cream by the patient and will assist the patient, if necessary. In addition, the patient will be scheduled to return for a safety evaluation approximately 1 week after completing treatment. The patient will be instructed to contact the site PI or designee if any unusual adverse events (AEs) occur during treatment or in the week after completing treatment. The patient will be scheduled to return to the MTF on Day 90 (± 14 days) days after starting treatment to determine whether all CL lesions have healed (as per CL standard of care). Those patients who cannot return to an MTF will be contacted by phone.

If at any time after completing treatment the lesions get worse or appear to be infected, the patient will be instructed to go to an MTF for possible treatment of AEs or alternative treatments for CL.

ELIGIBILITY:
Inclusion Criteria:

* Male or female military health care beneficiary of any age.
* Diagnosis of uncomplicated CL by having at least one lesion parasitologically confirmed by at least one of the following methods: 1) positive culture for promastigotes; 2) microscopic identification of amastigotes in stained lesion tissue; and/or 3) PCR assay performed either at the LDL, WRAIR or the Clinical Parasitology Service, CDC.
* Ability to comprehend and willingness to sign informed consent or give assent
* CL lesions in a location amenable to topical treatment
* Patient is willing to forgo other treatments for CL while on treatment program
* Females of childbearing potential must have a negative pregnancy test within 1 day of starting treatment and agree to use an acceptable method of birth control from start of treatment until 2 weeks after completing treatment

Exclusion Criteria:

* Clinically significant concomitant disease that would preclude the patient from completing treatment in the opinion of the treating physician.
* Clinical Evidence of mucosal involvement
* Known allergy to aminoglycosides
* Females who are pregnant or breastfeeding

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Aronson, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Military Treatment Facilities, Multiple Locations, Maryland

REFERENCES:
- [Background] Grogl M, Schuster BG, Ellis WY, Berman JD. Successful topical treatment of murine cutaneous leishmaniasis with a combination of paromomycin (Aminosidine) and gentamicin. J Parasitol. 1999 Apr;85(2):354-9. PMID 10219319